CLINICAL TRIAL: NCT05883462
Title: Prospective Trial of Paclitaxel-Coated Nasal Balloon for the Treatment of Recurrent Chronic Rhinosinusitis With or Without Nasal Polyps
Brief Title: Paclitaxel-Coated Nasal Balloon for the Treatment of Recurrent Chronic Rhinosinusitis With or Without Nasal Polyps (FIH)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Airiver Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESTORE-1
Record Dates: First submitted 2023-05-19; First posted 2023-06-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis
Keywords: recurrent, CRS with nasal polyps, CRS without nasal polyps
MeSH Terms: conditions — Recurrence | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm treated by Airiver Nasal DCB (Experimental): Subjects with recurrent symptomatic nasal obstruction will be treated by Airiver Nasal Drug Coated Balloon (DCB) Catheter at the index procedure. The balloon is coated with a paclitaxel drug (3.5ug/mm2).
  Interventions: Combination Product: Airiver Nasal Drug Coated Balloon (DCB) Catheter.

INTERVENTIONS:
Combination Product: Airiver Nasal Drug Coated Balloon (DCB) Catheter. — The balloon is coated with a paclitaxel drug (3.5ug/mm2).

SUMMARY:
It is a first in human (FIH) study to evaluate safety, and potential efficacy of Airiver Nasal DCB in the treatment of recurrent CRSwNP or CRSsNP.

Participants will receive AIRIVER Nasal drug-coated balloon treatment.

DETAILED DESCRIPTION:
Paclitaxel coated balloon is designed to offer both mechanical dilation of nasal obstruction and local drug effect for underlying inflammatory disorder and cell hyperplasia. It is hypothesized that Airiver Nasal drug-coated balloon (DCB) will improve patient outcome and as an adjunct to standard of care, will improve nasal patency than the standard of care alone. This is a prospective, single arm, first in human (FIH) study.

ELIGIBILITY:
Inclusion Criteria: Up to 45 CRS subjects with recurrent symptomatic nasal obstruction eligible for Airiver Nasal DCB treatment

1. Males or females, ≥18 years
2. Signed written informed consent
3. Recurrent, symptomatic CRS (with or without nasal polyps, with or without prior sinus surgery), have:

   * Moderate or severe nasal congestion/blockage/obstruction
   * AND decreased or loss of smell (hyposmia or anosmia),
   * Or rhinorrhea (anterior/posterior)

     * For recurrent CRSwNP:

       1. candidates for RESS or other treatment due to recurrent symptom, and endoscopically confirmed present with unilateral or bilateral polyps, and/or unilateral or bilateral mucosal disease confirmed by nasal endoscopy and/or CT
       2. bilateral sinonasal polyposis that despite prior treatment with systemic corticosteroids (SCS) anytime within the past 2 years; and/or had a medical contraindication / intolerance to SCS
       3. with or without Aspirin-Exacerbated Respiratory Disease (AERD)
     * For recurrent CRSsNP: refractory to optimal medical treatment and/or previous surgery with positive CT scan of the sinuses mucosal thickening and obstruction or positive nasal endoscopic finding (purulence or edema)
4. Acute Exacerbation of CRS (AECRS)
5. Subjects with comorbid asthma or COPD must be stable with no exacerbations (e.g., no emergency room visits, hospitalizations) for 6 months before the screening visit

Exclusion Criteria:

1. Pediatric CRS (PCRS)
2. Acute bacterial sinusitis (ABRS), acute rhinosinusitis (ARS), or mycetoma and invasive fungal sinusitis
3. Malignancy
4. Experienced a cerebrospinal fluid (CSF) leak in prior skull-based dehiscence
5. Symptomatic without positive CT findings or an asymptomatic
6. Subjects whose symptoms are too severe (eg, temperature >102.58F or extrasinus manifestations, such as orbital cellulitis; dental or facial or brain abscess; cavernous vein thrombosis; or altered mental status
7. Primary ciliary dyskinesia (PCD)
8. Unable to have nasal cavity examination due to septal deviation or spur. Participants who had a sinonasal or sinus surgery changing the lateral wall structure of the nose making impossible the evaluation of NP
9. Have evidence of significant baseline mucosal injury, ulceration, or erosion (eg, exposed cartilage, perforation) on baseline nasal examination
10. Purulent nasal infection, or upper respiratory tract infection within 2 weeks before the screening visit. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution
11. Allergy or hypersensitivity to any excipients and paclitaxel.
12. Patient has an inability to tolerate endoscopy
13. Suffering or recovering from COVID-19 (Fully recovered Covid-19 patients is not excluded)
14. Study subject has any disease or condition that interferes with safe completion of the study, such as severe COPD or severe asthma
15. Subjects with abnormal screening laboratory/imaging test results that compromise the ability to assess the benefits/risks (eg, abnormal ECG)
16. Pregnancy or planning on pregnant during the first 12 months of enrollment in the study
17. Life expectancy <1 year
18. Patient is currently enrolled in other current investigational studies. Participation in studies for products approved in the US are not considered investigational.
19. Lack of informed consent
20. Allergic granulomatous angiitis (Churg-Strauss syndrome), granulomatosis with polyangiitis (Wegener's granulomatosis), Young's syndrome, Kartagener's syndrome or other dyskinetic ciliary syndromes

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety: Freedom from major device related adverse events (MADE) post index procedure assessed by the proportion of subjects free from the primary safety event through 30 days. | 30 days
  Subjects failing any component of the primary safety endpoint will be considered a safety failure, and subjects who remain event free through 30 days will be considered safety successes. MADE is defined as: 1) Cerebrospinal fluid (CSF) leak, 2) Severe epistaxis (nasal bleeding) requiring intervention other than packing, 3) Eye complication requiring surgical treatment, 4) Paclitaxel related nasal mucosal disorder.
Primary efficacy: Freedom from target lesion reintervention due to recurrence of CRS without nasal polyposis or CRS with nasal polyposis (retuning to baseline symptoms or worse) through 6 months. | 6 months
  assessed by Kaplan-Meier survival analysis of the incidence of subjects free from symptom-driven TLR.

SECONDARY OUTCOMES:
Incidence of, and time to symptom-driven reintervention | 12 months
  assessed by Kaplan-Meier survival analysis of the incidence of subjects free from symptom-driven TLR
Change in patient reported 22-item Sino-Nasal Outcome Test (SNOT-22) from the baseline | 12 months
  Total SNOT 22 score is between 0 to 110. Higher scores indicate worse rhinosinusitis.
Change in Lund-Kennedy Endoscopic Scores from the baseline | 12 months
  The scores range is from 0 to 20. Higher scores indicate worse observed disease.
Change in Lund-Mackay computed tomography (LMK-CT) score from the baseline | 12 months.
  The score range is from 0 to 24. Higher scores indicate worse disease severity.
Change of Health-related quality -of- life (HRQL) from the baseline (Euro-QOL-5D questionnaire) | 12 months
  The EQ-5D essentially consists of 2 parts: the EQ-5D descriptive system and the EQ VAS. The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a vertical VAS. The EQ VAS 'thermometer' has scales of 100 (Best imaginable health state) at the top and 0 (Worst imaginable health state) at the bottom.
Change in sense of smell using the University of Pennsylvania Smell Identification Test (UPSIT) from the baseline | 12 months
  The score range is between 0-40. Higher scores indicate better smell function.
Clinical pharmacokinetics of paclitaxel in 15 subjects | 10 days
  Blood samples will be collected at baseline and post procedure at pre-designated time points and assessed for plasma paclitaxel concentrations.
Change in Asthma Control Questionnaire-6 (ACQ-5) Scores from baseline for subjects with comorbid asthma | 12 months
  A score of 0-6 is assigned to values for each criterion. The total ACQ score is the mean value calculated after adding the individual scores for each criterion. In general, patients with a score below 1.0 are likely to have adequately controlled asthma, above 1.0 their asthma is not likely to be well-controlled.
Nasal DCB performance evaluation in index procedures | one day
  Device Performance will be assessed using a rating scale (1-5) to evaluate seven aspects of the test article. Higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Coral Leticia Benítez Insaurralde, MD, Principal Investigator — Sanatorio Americano Hospital
Locations (1):
- Sanatorio Americano Hospital, Asunción, Paraguay